CLINICAL TRIAL: NCT04804618
Title: Exploring Research on Early Warning Indicators of Protein in Patients With Mild Cognitive Impairment and Alzheimer's Disease
Brief Title: Proteomics Study of Mild Cognitive Impairment and Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: Guangzhou Cadre Health Management Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: AD2020
Record Dates: First submitted 2021-02-20; First posted 2021-03-18 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Alzheimer Disease, Early Onset; Protein; Disease
Keywords: Alzheimer Disease; biomarker; protein
MeSH Terms: conditions — Alzheimer Disease; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All biological specimens (including blood, feces, urine, saliva and tongue coating) will be stored in the biological resource center of the our research centers after written informed consent obtained from all subjects who voluntarily participated in this clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy control group: aged ≥55 years old, no dementia, MCI or no family history of AD.
- Alzheimer's disease high-risk group: aged ≥55 years old, immediate family members of AD patients
- Alzheimer's disease group: aged ≥55 years old, diagnosed as AD patients
- Mild cognitive impairment group: patients ≥55 years of age, diagnosed with MCI

SUMMARY:
This study intends to adopt standardized and rigorous cross-sectional research, collect biological specimens (including blood, feces, urine, saliva and tongue coating) from eligible subjects, and use liquid chromatography/mass spectrometry (LC-MS/MS) technology to explore early warning indicators of protein in patients with mild cognitive impairment and Alzheimer's disease

DETAILED DESCRIPTION:
The problem of population aging is getting worse, the prevalence of senile dementia is increasing, and Alzheimer's disease (AD) is the most common type of dementia. There is no effective treatment for AD. Most interventions can only alleviate the condition and delay the development. Therefore, early diagnosis and prevention of AD are extremely important. However, the current diagnostic measures are not suitable for clinical promotion due to their traumatic nature, so there is an urgent need for a more suitable clinical early identification and diagnosis method. Proteomics research technology is the leading research technology in China. It can be applied to research on disease markers, pathogenesis, and drug target discovery.

Therefore, this study intends to adopt standardized and rigorous cross-sectional research, collect biological specimens (including blood, feces, urine, saliva and tongue coating) from eligible subjects, and use liquid chromatography/mass spectrometry (LC-MS/MS) technology to explore early warning indicators of protein in patients with mild cognitive impairment and Alzheimer's disease

ELIGIBILITY:
Inclusion Criteria:

1. Older than 55-year-old，male or female.
2. patients meet the diagnosis of mild cognitive impairment (MCI) or Alzheimer's disease(AD) or whose family members were diagnoed with AD
3. Complete self-rating scale for memory impairment (AD-8 scale)
4. Those who agree to participate in clinical research and sign informed consent.

Exclusion Criteria:

1. Patients with acute cardiovascular and cerebrovascular diseases, acute infections (pneumonia, urinary tract infection, oral infection, digestive tract infection), severe renal dysfunction, and uremia;
2. Pregnant or lactating women;

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: From March 2021 to March 2022，people who finish the cognitive examination at Guangdong Provincial Hospital of Chinese Medicine and the Guangzhou Cadre Health Management Center would be this study population. All the eligible participants will be follow up every year until 2026.
Sampling Method: Probability Sample
Enrollment: 650 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the protein expression profile of urine and saliva | An Average of 1 year
  Proteomic expression of urine and saliva in each group will be tested use Protein liquid chromatography/mass spectrometry detection.

SECONDARY OUTCOMES:
Change of the cognitive function every year | An Average of 1 year
  Mini-mental State Examination (MMSE) score for the the cognitive function assessment. The total score in MMSE ranges from 0 to 30, and higher scores indicate better cognition.
Changes in plasma protein expression profile every year | An Average of 1 year
  Proteomic expression of plasma in each group will be tested use Protein liquid chromatography/mass spectrometry detection.
Variation characteristics of gut microbiome every year | An Average of 1 year
  Bacterial genomic DNA was extracted from faecal and tongue coating samples of each group using 16S RNA sequencing and analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Province Hospital of Tradtional Chinese Medicine, Guangzhou, Guangdong, China